CLINICAL TRIAL: NCT00240123
Title: Effect of Diphenhydramine Sedation During Endoscopic Retrograde Cholangio-pancreatography (ERCP) or Endoscopic Ultrasound (EUS)
Brief Title: Effect of Benadryl Sedation During ERCP or EUS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10454
Record Dates: First submitted 2005-09-13; First posted 2005-10-17 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Gallbladder Disease; Gallstones; Pancreatitis; Abdominal Pain; Jaundice
Keywords: ERCP; EUS
MeSH Terms: conditions — Gallbladder Diseases; Gallstones; Pancreatitis; Abdominal Pain; Jaundice

INTERVENTIONS:
Drug: Benadryl versus Placebo

SUMMARY:
The purpose of the study is to determine if adding Benadryl improves sedation for patients scheduled to undergo ERCP or EUS procedures.

DETAILED DESCRIPTION:
The usual sedatives used for endoscopy are meperidine (Demerol) and midazolam (Versed). Benadryl (Diphenhydramine) is often used in addition to these medications in an effort to improve sedation. There is little published information regarding the use of diphenhydramine in conscious sedation. It is recognized that certain patients have features that predict difficult sedation such as prescription sedative use or heavy alcohol use. In addition, prolonged procedures like ERCP and EUS require higher doses of sedatives. Diphenhydramine may improve the quality of sedation in patients undergoing endoscopic retrograde cholangio-pancreatography (ERCP) or endoscopic ultrasound (EUS) procedures. You are being asked to participate because you are already scheduled to undergo one of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age who present for outpatient ERCP or EUS at Strong Memorial Hospital Endoscopy Center will be included

Exclusion Criteria:

* Allergy to diphenhydramine, narrow angle glaucoma, or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Study Completion 2007-07

PRIMARY OUTCOMES:
Recovery score

SECONDARY OUTCOMES:
Quality of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Maliakkal, MD, Principal Investigator — University of Rochester Medical Center, Digestive and Liver Disease Unit